CLINICAL TRIAL: NCT06220370
Title: PATH Study: People With Injecting Related Infections: Assessing Treatment Outcomes for Those Who Are Hospitalised.
Acronym: PATH
Status: Not yet recruiting | Type: Observational
Sponsor: Kirby Institute (Other Government)
Responsible Party: Sponsor
Other Study IDs: PATH
Record Dates: First submitted 2024-01-14; First posted 2024-01-23 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-01

CONDITIONS: Invasive Fungal Infections; Invasive Bacterial Infection; Injection Site Infection; Infection, Bacterial; Infection, Fungal; Infection, Soft Tissue
Keywords: Antimicrobial therapy; Patient-directed discharge; Injection-related infectious diseases
MeSH Terms: conditions — Invasive Fungal Infections; Bacterial Infections; Mycoses; Soft Tissue Infections | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational — There is no clinical intervention as part of this study. Participants will receive treatment as per their clinical treating team.

SUMMARY:
We seek to characterise the burden and outcomes of and understand the current experience of people who inject drugs admitted to hospital with invasive injecting-related infections, in order to implement and evaluate strategies to improve completion of therapy and reduce patient-directed discharges, with ultimate benefit to the patient and health service.

DETAILED DESCRIPTION:
This study will be conducted as a prospective, observational cohort study of adults admitted with invasive bacterial and fungal infectious diseases. This study will be conducted at multiple hospitals in Australia.

Participants will be invited for Screening whilst they are inpatients of the hospital. Participants will be screened for history of injection drug use in the last 6 months and presence of an invasive bacterial or fungal infection.

Eligible participants will be treated through standard of care with the applicable treatment. All participants will commence antimicrobial treatment whilst they are inpatients. For participants who are discharged before planned treatment completion, a hospital discharge visit (Early Discharge Electronic Case Report Form [eCRF]) will be conducted. Following the end of treatment, participants will be reviewed at 6, 12 and 48-weeks post-enrolment. At follow-up visits, behavioural surveys, health-related quality of life, and experiences with hospital care will be assessed.

Individual patient involvement will include four visits over a 12-month period.

The duration of the study is anticipated to be 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Have voluntarily signed the informed consent form,
2. 18 years of age or older,
3. Injected drugs within the last 6 months,
4. Admitted to hospital with invasive bacterial or fungal infection, a. Examples of invasive infection include: bloodstream infection, bone and joint infection (osteomyelitis, septic arthritis, discitis), central nervous system infection (epidural abscess, meningitis), deep abscess (i.e., brain, liver, muscle, spleen), endovascular infection (infective endocarditis, septic thrombophlebitis, mycotic aneurysm, septic embolism), skin or soft tissue infection (necrotising fasciitis, myositis),

Exclusion Criteria:

1) Is unable or unwilling to provide informed consent or abide by the requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be conducted as a prospective, observational cohort study of adults admitted with invasive bacterial and fungal infectious diseases. This study will be conducted at multiple hospitals in Australia.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2029-03-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
primary outcome | 5 years
  To evaluate the proportion electing for, and factors associated with, patient-directed discharge among PWID admitted for management of invasive IRID.

IPD SHARING:
Plan to Share IPD: No